CLINICAL TRIAL: NCT04062084
Title: Study of Multifunctional Cataract-assisted Retractor in Complicated Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: xuwen2017-034
Record Dates: First submitted 2019-07-31; First posted 2019-08-20 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2020-12

CONDITIONS: Subluxation of Lens; Surgical Instruments，Cataract
MeSH Terms: conditions — Lens Subluxation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multifunctional Cataract-assisted Retractor (Experimental): Patients undergoing cataract with lens subluxation surgery with Multifunctional cataract-assisted retractor
  Interventions: Device: Multifunctional Cataract-assisted Retractor
- Capsule Retractor (Experimental): Patients undergoing cataract with lens subluxation surgery with traditional capsule retractor
  Interventions: Device: Multifunctional Cataract-assisted Retractor

INTERVENTIONS:
Device: Multifunctional Cataract-assisted Retractor — Multifunctional Cataract-assisted retractor operation for cataract with subluxation of lens

SUMMARY:
To compare the safety and efficacy of a new multi-functional cataract-assisted surgical instrument with that of traditional cataract-assisted surgical instrument in cataract surgery with subluxation of lens.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of lens subluxation.
* Patients need to undergo lens subluxation surgery

Exclusion Criteria:

* Active intraocular inflammation
* The intraocular pressure (IOP) was higher than 25 mmHg
* The endothelial cell count (ECC) was less than 1,200 cells/mm2
* Combined with other eye diseases
* Combined with other serious systemic diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Surgical success rate | through study completion, an average of 1 year
  Surgical success rate of operation with different retractor

SECONDARY OUTCOMES:
Successful implantation rate of intraocular lens | through study completion, an average of 1 year
  implantation rate of intraocular lens with different retractor
Visual function | 1day postoperation，1 week，1 month， 3month postoperation
  Best corrected visual acuity (BCVA) measured using a decimal chart Best corrected visual acuity (BCVA) measured using a decimal chart
intraocular pressure | 1 day, 1 week, 1 month, and 3 month postoperation
  intraocular pressure
endothelial cell count | 1 week, 1 month, and 3 month postoperation
  endothelial cell count

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No